CLINICAL TRIAL: NCT03694210
Title: Prospective, Trial Evaluating the Safety and Effectiveness of the Interscope Endorotor® System for Direct Endoscopic Necrosectomy of Walled Off Pancreatic Necrosis
Brief Title: EndoRotor DEN (Direct Endoscopic Necrosectomy)Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Interscope, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0047
Record Dates: First submitted 2018-09-26; First posted 2018-10-03 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Acute Pancreatic Necrosis; Acute Pancreatitis; Necrotizing Pancreatitis
Keywords: Direct Endoscopic Necrosectomy; Walled Off Necrosis; Walled Off Pancreatic Necrosis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Intervention Model Description: A prospective, single arm, open label, multi-center, trial to evaluate the safety and effectiveness of the Interscope EndoRotor® Resection System in subjects requiring direct endoscopic necrosectomy with walled off pancreatic necrosis (WOPN).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EndoRotor Therapy (Experimental): Physicians will perform direct endoscopic necrosectomy using the EndoRotor in patients with walled off necrosis.
  Interventions: Device: EndoRotor Therapy

INTERVENTIONS:
Device: EndoRotor Therapy — To evaluate the EndoRotor's ability to safely remove non-viable/necrotic tissue for direct endoscopic necrosectomy in patients with walled off pancreatic necrosis.

SUMMARY:
A prospective, single arm, open label, multi-center, trial to evaluate the safety and effectiveness of the Interscope EndoRotor® Resection System in subjects requiring direct endoscopic necrosectomy (DEN) with walled off pancreatic necrosis (WOPN).

DETAILED DESCRIPTION:
A prospective, single arm, open label, multi-center, trial to evaluate the safety and effectiveness of the Interscope EndoRotor® Resection System in subjects requiring direct endoscopic necrosectomy with walled off pancreatic necrosis (WOPN). Total enrollment 30 subjects with at least 15 enrolled in the US.

Subjects will be debrided with the EndoRotor either at the time of stent placement or post placement at Investigator's discretion with a maximum of 4 EndoRotor procedures. A minimum of 2 days is required between each EndoRotor procedure and all procedures need to be completed within a 14 (+7/-0) day period. Follow up is completed 21 (+/- 7) days after last EndoRotor debridement procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are >22; inclusive of males and females.
2. Patients with symptomatic pancreatic necrosis due to acute pancreatitis that have an indication to undergo endoscopic necrosectomy after having undergone EUS-guided drainage
3. Imaging suggestive of greater than or equal to 30% necrotic material
4. Walled off pancreatic necrosis size ≥6 cm and ≤22cm
5. Subject can tolerate repeated endoscopic procedures
6. Subject capable of giving informed consent.
7. Subjects with the ability to understand the requirements of the study, who have provided written informed consent, and who are willing and able to return for the required follow-up assessments through 21 (+/- 7) days, as indicated.

Exclusion Criteria:

1. Subject unable to give informed consent.
2. Subject is unwilling to return for repeated endoscopies.
3. Documented Pseudoaneurysm > 1cm within the WOPN
4. Intervening gastric varices or unavoidable blood vessels within the access tract (visible using endoscopy or endoscopic ultrasound).
5. Dual antiplatelet therapy or therapeutic anticoagulation that cannot be withheld for the procedure
6. Any condition that in the opinion of the investigator would create an unsafe clinical situation that would not allow the patient to safely undergo an endoscopic procedure (lack of medical clearance).
7. Pregnant or lactating women or women of childbearing potential who do not employ a reliable method of contraception as judged by the Investigator, and/or are not willing to use reliable contraception for the duration of study participation.
8. Patient is known to be currently enrolled in another investigational trial that could interfere with the endpoint analyses of this trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bruno, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (10):
- United States (7):
  - Benjamin Tharian, Little Rock, Arkansas
  - Stanford University Medical Center, Palo Alto, California
  - California Pacific Medical Center - Sutter Health, San Francisco, California
  - University of Chicago Department of Medicine, Chicago, Illinois
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Arvin Trindade, Queens, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- Germany (2):
  - University of Frankfurt Medicine, Frankfurt
  - Interdisciplinary Clinic for Endoscopy - TU Munich, München
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stassen PMC, de Jonge PJF, Bruno MJ, Koch AD, Trindade AJ, Benias PC, Sejpal DV, Siddiqui UD, Chapman CG, Villa E, Tharian B, Inamdar S, Hwang JH, Barakat MT, Andalib I, Gaidhane M, Sarkar A, Shahid H, Tyberg A, Binmoeller K, Watson RR, Nett A, Schlag C, Abdelhafez M, Friedrich-Rust M, Schlachterman A, Chiang AL, Loren D, Kowalski T, Kahaleh M. Safety and efficacy of a novel resection system for direct endoscopic necrosectomy of walled-off pancreas necrosis: a prospective, international, multicenter trial. Gastrointest Endosc. 2022 Mar;95(3):471-479. doi: 10.1016/j.gie.2021.09.025. Epub 2021 Sep 22. PMID 34562471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Dates: November 2018 to August 2019
Period: Overall Study
Arm/Group | EndoRotor Therapy
Started (37 patients were screened, 7 were screen failures, 30 were enrolled and treated.) | 37
Completed (1 subject passed away just prior to completing the study but all analysis points were collected prior to this.) | 29
Not Completed | 8
Not completed — Death | 1
Not completed — Screen Failure | 7

BASELINE CHARACTERISTICS:
Population: 30 subjects were enrolled and treated. 1 subject did not complete follow-up (21 days following the final necrosectomy) as they expired; however, all data points were collected for analysis prior to this.
Arm/Group | EndoRotor Therapy
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  Netherlands | 2
  United States | 23
  Germany | 5
Cause of Pancreatitis [Count of Participants; unit: Participants]
  Gallstone/biliary | 18
  Alcohol | 5
  Unknown Cause | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Device Related Complications
Description: The primary endpoint of this study is the freedom from major device related complications. The safety endpoint will include an assessment of the safety of the EndoRotor when performing endoscopic necrosectomy. For the purpose of this study, the safety evaluation shall include complications associated with endoscopic necrosectomy through the 21 (+/-7) day follow-up period. Potential endoscopic complications include perforation and bleeding.
Time Frame: 21 +/- 7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRotor Therapy
Number analyzed (Participants) | 30
Participants | 0

2. Secondary Outcome: Effectiveness: Number of Participants With at Least 70% of Necrotic Debris Removed
Description: Successful clearance of necrosis in the collection being treated during direct endoscopic necrosectomy where success is defined as at least 70% of the necrotic debris in the collection being treated is removed based on CT evaluation of the cavity at the 21 (+/-7) day follow up visit.
Time Frame: 21 +/- 7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | EndoRotor Therapy
Number analyzed (Participants) | 30
Participants | 29

3. Secondary Outcome: Mean Total Procedure Time to Achieve at Least 70% Reduction in Necrosis
Description: Assessment of total procedure time to achieve clearance of necrosis for all procedures.
  Total procedure time is measured from scope-in to scope-out. EndoRotor time is measured from the start of EndoRotor use to the end of EndoRotor use.
Time Frame: Completion of all necrosectomy procedures per patient
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | EndoRotor Therapy
Number analyzed (Participants) | 30
Minutes
  Total Procedure Time | 117 (50)
  EndoRotor Time | 71 (37)

4. Secondary Outcome: Adequacy of Procedural Debridement: Mean Percent Necrotic Material Removed From the WOPN Cavity Per Procedure.
Description: At the completion of each necrosectomy procedure the Investigator will visually inspect the WOPN cavity endoscopically and estimate the percent of necrosis that was removed from the cavity using EndoRotor. For each procedure, the initial amount of necrosis in the WOPN cavity is considered 100%.
Time Frame: This outcome was assessed at the completion each necrosectomy procedure per participant. At the completion of all necrosectomy procedures for all participants, an overall mean percent necrotic material removed from the WOPN per procedure was calculated.
Measure: Mean (Standard Deviation); unit: % Necrosis removed for all procedures
Arm/Group | EndoRotor Therapy
Number analyzed (Participants) | 30
% Necrosis removed for all procedures | 60 (33)

5. Secondary Outcome: Mean Number of Necrosectomy Procedures Required Per Participant to Achieve at Least 70% Reduction in Necrosis.
Description: The total number of necrosectomy procedures required per participant to achieve at least 70% reduction in necrosis from the WOPN will be assessed.
Time Frame: This outcome was assessed at completion of all necrosectomy procedures per participant. After completion of all necrosectomy procedures in all participants the overall mean number of procedures to achieve at least 70% reduction in necrosis was calculated.
Measure: Mean (Standard Deviation); unit: Procedures
Arm/Group | EndoRotor Therapy
Number analyzed (Participants) | 30
Procedures | 2 (2)

6. Secondary Outcome: Mean Length of Hospital Stay Per Participant
Description: The total length of hospital stay per participant measured in days, from the date of the index necrosectomy procedure to the date of discharge.
Time Frame: At patient discharge from hospital
Population: Patients with outpatient visits were assigned 0.5 days conservatively
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EndoRotor Therapy
Number analyzed (Participants) | 30
Days | 18 (25)

7. Secondary Outcome: Quality of Life - Short Form 36-Item Health Survey Version 1 (SF-36v1), Physical & Emotional Composite Score
Description: The SF-36v1 questionnaire measures functional health and well-being from a patient's point of view. The questionnaire assess eight health domains including: Physical Functioning, Role Limitations due to Physical Health, Role Limitations due to Emotional Problems, Energy/Fatigue, Emotional Well Being, Social Functioning, Pain, and General Health.
  Participants were asked to complete the questionnaire at the Baseline Visit and then again at the 21 Day Post Necrosectomy Follow-up Visit. The results of the questionnaire from the 21 Day Post Necrosectomy Follow-up Visit were then compared to those of Baseline for improvement.
  Numeric scores for each health domain are reported on a scale of 0-100 with improvement demonstrated by a higher score than baseline. Statistically significant improvement is denoted by differences in Baseline and 21 Day Follow-up Visit scores that have a p-value < 0.05.
Time Frame: 21 +/- 7 Days
Population: All participants who had a completed SF-36v1 Questionnaire at both Baseline and the 21 Day Follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline SF-36v1 Score: Baseline SF-36v1 results for 8 domains
- 21 Day Post Necrosectomy SF-36v1 Score: 21 Day Post Necrosectomy SF-36v1 results for 8 domains
Arm/Group | Baseline SF-36v1 Score | 21 Day Post Necrosectomy SF-36v1 Score
Number analyzed (Participants) | 24 | 24
score on a scale
  Physical Functioning | 36.0 (30.8) | 57.3 (30.8)
  Role Limitations due to Physical Health | 11.4 (28.5) | 25.0 (37.6)
  Role Limitations due to Emotional Problems | 27.8 (41.3) | 51.4 (48.1)
  Energy / Fatigue | 27.9 (22.0) | 36.7 (23.2)
  Emotional Well Being | 60.7 (19.7) | 68.3 (18.9)
  Social Functioning | 51.6 (32.6) | 56.3 (26.6)
  Pain | 31.4 (28.4) | 56.0 (30.1)
  General Health | 47.8 (15.9) | 53.8 (15.3)
Statistical Analysis 1: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; Physical Functioning: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.0011, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0
Statistical Analysis 2: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; Role Limitations due to Physical Health: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.1152, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0
Statistical Analysis 3: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; Role Limitations due to Emotional Problems: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.0552, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0
Statistical Analysis 4: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; Energy/Fatigue: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.039, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0
Statistical Analysis 5: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; Emotional Well Being: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.0223, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0
Statistical Analysis 6: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; Social Functioning: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.4664, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0
Statistical Analysis 7: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; Pain: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.0001, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0
Statistical Analysis 8: Comparison: Baseline SF-36v1 Score vs 21 Day Post Necrosectomy SF-36v1 Score; General Health: 21 Day Post Necrosectomy SF-36v1 Score is compared to Baseline score for improvement; Test type: Superiority; p = 0.0639, Wilcoxon Signed Rank Test — p-values of <0.05 are considered significant; Mean Difference (Net) = 0

ADVERSE EVENTS:
Time Frame: Adverse Events were captured from Index Procedure through 21 day Follow-up
Arm/Group | EndoRotor Therapy
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 9/30
Other Adverse Events (participants affected / at risk) | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoRotor Therapy (N=30)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) — Moderate severity, not related to device, not related to procedure
Hematemesis (Gastrointestinal disorders) | 1 (1) — Moderate severity, not related to device, not related to procedure
Sepsis (Infections and infestations) | 1 (1) — Moderate severity, not related to device, not related to procedure
Cholestasis (Hepatobiliary disorders) | 1 (1) — Moderate severity, not related to device, not related to procedure
Gastrointestinal Bleed (Gastrointestinal disorders) | 2 (2) — Event 1: Severe severity, not related to device, possible relationship to procedure Event 2: Moderate severity, not related to device, possible relationship to procedure
Pneumoperitoneum (Surgical and medical procedures) | 1 (1) — Mild severity, not related to device, possible relationship to procedure
Multiple Organ Failure Syndrome (General disorders) | 1 (1) — Severe severity, not related to device, not related to procedure. Patient later deceased
Pancreatitis (Hepatobiliary disorders) | 1 (1) — Severe severity, not related to device, not related to procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoRotor Therapy (N=30)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Moderate severity, not related to device, not related to procedure
Bacteremia (Infections and infestations) | 1 (1) — Moderate severity, not related to device, not related to procedure
Colitis (Gastrointestinal disorders) | 1 (1) — Mild severity, not related to device, not related to procedure
Diarrhea (Gastrointestinal disorders) | 1 (1) — Mild severity, no related to device, not related to procedure
Esophageal Candidiasis (Gastrointestinal disorders) | 1 (1) — Moderate severity, not related to device, not related to procedure
Pyrexia (General disorders) | 1 (1) — Moderate severity, not related to device, not related to procedure
Clostridium Difficile Infection (Infections and infestations) | 1 (1) — Moderate severity, not related to device, not related to procedure
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) — Mild severity, not related to device, not related to procedure
Insomnia (Nervous system disorders) | 1 (1) — Mild severity, not related to device, not related to procedure
Device Dislocation (LAMS dislodgement) (Product Issues) | 1 (1) — Mild severity, not related to device, definitely related to procedure
Anemia (Vascular disorders) | 1 (1) — Moderate severity, not related to device possible relationship to procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty days before publication submission PI shall submit to Sponsor for review and comment. PI will consider comments, but is not obligated to incorporate suggestions. Publication shall acknowledge Sponsor contributions as appropriate. Investigator agrees that first publication of results shall be a joint, multicenter publication, with the investigators and the institutions from all appropriate sites contributing data, analyses and comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT03694210/Prot_SAP_000.pdf